CLINICAL TRIAL: NCT00333320
Title: Positive Effect of Ischemic Postconditioning During Acute Myocardial Infarction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POSTCONDITIONING; SFC-2006-02
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; postconditioning; coronary reserve; ejection fraction
MeSH Terms: interventions — Ischemic Postconditioning; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- - Control (Placebo Comparator)
  Interventions: Procedure: Control group
- -postconditioning group (Experimental)
  Interventions: Procedure: postconditioning

INTERVENTIONS:
Procedure: postconditioning — patients were treated by repeated cycles of cycles of reperfusion/ischemia at the end of the procedure within the first minute after reperfusion
  Arms: -postconditioning group
Procedure: Control group — Percutaneous coronary interventions were performed following international guidelines. No additional intervention was performed in the control group.
  Arms: - Control

SUMMARY:
The purpose of this study is to determine whether brief periods of ischemia performed just at the time of reperfusion -postconditioning- can reduce coronary endothelial dysfunction and infarct size in humans

DETAILED DESCRIPTION:
Desobstruction of the culprit artery after acute myocardial infarction allows to reduce the consequences of prolonged ischemia. However, it is now clearly established that reperfusion induces by itself severe myocardial injuries. Postconditioning has been described as an adaptive response triggered by a brief ischemia applied after a prolonged coronary occlusion. Several teams have reported that ischemia/reperfusion cycles allow to reduce infarct size in experimental models.

Different pathophysiological processes have been proposed to explain the beneficial effect of postconditioning. It has been reported that postconditioning reduces the inflammatory response, and activates cardioprotective signaling pathways (Akt, eNOS, p70S6K). In addition, an improvement of the endothelial function has been reported.

This controlled trial aim to study the potential beneficial effect of postconditioning in patients with acute myocardial infarction. Forty six patients will be included in the study and the culprit artery will be reoccluded three times for 1 minutes after desobstruction in one of the both groups after randomization of the patients.

The evaluation will be focused on the comparison of the coronary reserve after intracoronary adenosine injection. In addition, additional parameters will be used to study the effect of postconditioning on post-ischemic endothelial dysfunction: frequencies of low reflow and slow reflow situation, myocardial blush and regression of ST elevation. The effect of postconditioning on the left ventricular systolic function will be studied by Doppler tissue imaging and RMN.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction (<6 hours)
* Occlusion of a major coronary vessel

Exclusion Criteria:

* History of previous myocardial infarction
* History of Coronary Artery Bypass Grafting
* Need for Coronary Artery Bypass Grafting
* Stenosis not eligible for angioplasty
* Limited ischemic area
* Cardiogenic shock
* Interventricular septum rupture
* Mitral regurgitation>2
* Ventricular tachycardia
* Atrioventricular block class II and III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
coronary reserve after intracoronary adenosine injection | Immediately after the postconditioning procedure

SECONDARY OUTCOMES:
frequencies of low reflow and slow reflow situation | after postconditioning
regression of ST elevation | 1h and 24h after postconditioning
left ventricular systolic function by Doppler tissue imaging (DAY 1 and 6) | day 1 and 6
left ventricular systolic function by RMN | day 8-12
myocardial blush | after postconditioning

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Le Corvoisier, MD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Henri Mondor University Hospital, Créteil, France